CLINICAL TRIAL: NCT01438229
Title: Ablation-induced Renal Sympathetic Denervation Trial
Brief Title: Safety and Efficacy Study of Renal Artery Ablation in Resistant Hypertension Patients
Acronym: EnligHTN-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CI-10-045-ID-HT; Arsenal (Other: St Jude Medical)
Record Dates: First submitted 2011-09-19; First posted 2011-09-22 (Estimated); Results first posted 2015-05-21 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Hypertension
Keywords: Catheter-based renal artery ablation; Hypertension; Resistant to Conventional Therapy
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- renal artery ablation (Experimental): Catheter-based RF ablation in renal artery
  Interventions: Device: St. Jude Medical renal artery ablation system: RF ablation generator (IBI 1500T11.5) and Renal artery ablation catheter (DS3D001, DS3D002)

INTERVENTIONS:
Device: St. Jude Medical renal artery ablation system: RF ablation generator (IBI 1500T11.5) and Renal artery ablation catheter (DS3D001, DS3D002) — Catheter-based RF ablation in renal artery

SUMMARY:
This is a prospective, multicenter, feasibility study on the safety and efficacy of renal denervation in patients with resistant hypertension.

DETAILED DESCRIPTION:
Demonstrate the safety and efficacy of the St. Jude Medical Radiofrequency (RF) Renal Denervation System in the treatment of patients with resistant hypertension.

Safety Marker

* All adverse events

Efficacy Marker

* Office blood pressure

ELIGIBILITY:
Inclusion Criteria:

* Office systolic blood pressure that remains ≥160 mmHg (≥150 mmHg for patient with type 2 diabetes) despite the stable use of ≥3 antihypertensive medications concurrently at maximally tolerated doses, of which one is a diuretic, for a minimum of 14 days prior to enrollment
* Age ≥18 and ≤80 years old
* Able and willing to provide written informed consent to participate in the study
* Able and willing to comply with the required follow-up schedule

Exclusion Criteria:

* Prior renal artery intervention (balloon angioplasty or stenting)
* Evidence of renal artery atherosclerosis (defined as a stenotic severity of >30%) in either renal artery
* Multiple main renal arteries in either kidney
* Main renal arteries <4 mm in diameter or <20 mm in length
* eGFR of <45 mL/min per 1.73 m2 using the MDRD formula
* Type 1 diabetes
* Renovascular hypertension or hypertension secondary to other renal disorders (glomerulonephritis, polycystic kidney disease, end-stage renal failure)
* Others

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2011-10; Primary Completion 2012-09 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vasilias Papademetriou, MD, Principal Investigator — First Cardioligy Clinic, Hippokration Hospital, University of Athens, Greece; Konstantinos Tsioufis, MD, Principal Investigator — First Cardioligy Clinic, Hippokration Hospital, University of Athens, Greece; Stephen Worthley, MD, Principal Investigator — Cardiovascular Investigation Unit, Royal Adelaide Hospital, Adelaide, Australia; Ian Meredith, MD, Principal Investigator — Monash Medical Centre, Melbourne, Australia; Derek Chew, MD, Principal Investigator — Flinders Medical Centre, Adelaide, AUSTRALIA
Locations (4):
- Australia (3):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Adelaide, South Australia
  - Monash Medical Centre, Melbourne, Victoria
- Hippokration Hospital, Athens, Greece

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Renal Artery Ablation
Started | 47
Excluded Due to Renal Artery Anatomy | 1
Underwent Procedure | 46
Completed | 44
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: Subjects completing renal artery ablation procedure
Arm/Group | Renal Artery Ablation
Number analyzed (Participants) | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 31
Race/Ethnicity, Customized [Number; unit: participants]
  White | 45
  Other | 1
Region of Enrollment [Number; unit: participants]
  Greece | 20
  Australia | 26
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 32 (5)
Coronary Artery Disease [Number; unit: participants]
  Yes | 9
  No | 37
Hyperlipidemia [Number; unit: participants]
  Yes | 27
  No | 19
Type II Diabetes Mellitus [Number; unit: participants]
  Yes | 15
  No | 31
Sleep Apnea [Number; unit: participants]
  Yes | 14
  No | 32
eGFR [Mean (Standard Deviation); unit: mL/min/1.73m^2] | 87 (19)
Serum Creatinine [Mean (Standard Deviation); unit: mmol/L] | 78 (17)
Cystatin C [Mean (Standard Deviation); unit: mg/L] | 1.1 (0.3)
Urine Albumin-to-Creatinine Ration [Mean (Standard Deviation); unit: mg/g] | 167.6 (493)
Number of Anti-Hypertensive Medications [Mean (Standard Deviation); unit: medications] | 4.7 (1.0)
Office Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 176 (16)
Office Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 96 (14)
Heart Rate [Mean (Standard Deviation); unit: beats per minute] | 71 (12)

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: All device or procedure related adverse events
Time Frame: 24 months
Population: All subjects receiving renal artery ablation procedure
Measure: Number; unit: percentage of participants
Arm/Group | Renal Artery Ablation
Number analyzed (Participants) | 46
percentage of participants | 47.8

2. Primary Outcome: Office Systolic Blood Pressure Change
Time Frame: Baseline to 6 months
Population: Subjects with both baseline and 6M follow up office blood pressure measurements
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Artery Ablation
Number analyzed (Participants) | 45
mmHg | -26 (25)
Statistical Analysis 1: Comparison: Renal Artery Ablation; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

3. Other Pre Specified Outcome: Office Diastolic BP Change
Time Frame: Baseline to 6M
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Artery Ablation
Number analyzed (Participants) | 45
mmHg | -10.5 (12.2)

4. Other Pre Specified Outcome: Office Systolic BP Change
Time Frame: Baseline to 12M
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Artery Ablation
Number analyzed (Participants) | 45
mmHg | -26.7 (20.9)

5. Other Pre Specified Outcome: Office Systolic BP Change
Time Frame: Baseline to 18 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Artery Ablation
Number analyzed (Participants) | 44
mmHg | -24.1 (20.4)

6. Other Pre Specified Outcome: Office Systolic BP Change
Time Frame: Baseline to 24 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Artery Ablation
Number analyzed (Participants) | 44
mmHg | -29.1 (26.1)

7. Other Pre Specified Outcome: Office Diastolic BP Change
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Artery Ablation
Number analyzed (Participants) | 45
mmHg | -10.7 (12.6)

8. Other Pre Specified Outcome: Office Diastolic BP Change
Time Frame: Baseline to 18 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Artery Ablation
Number analyzed (Participants) | 44
mmHg | -10.1 (11.9)

9. Other Pre Specified Outcome: Office Diastolic BP Change
Time Frame: Baseline to 24 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Artery Ablation
Number analyzed (Participants) | 44
mmHg | -13.3 (14.8)

10. Other Pre Specified Outcome: 24hr Ambulatory Systolic BP Change
Description: Average of readings taken every half hour during the course of a 24hr period wearing the ambulatory blood pressure monitor. Includes only subjects who completed the test at both baseline and follow up. If a subject refused to wear the monitor they were excluded.
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Artery Ablation
Number analyzed (Participants) | 44
mmHg | -10.3 (13.9)

11. Other Pre Specified Outcome: 24hr Ambulatory Systolic BP Change
Description: as for outcome 10
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Artery Ablation
Number analyzed (Participants) | 35
mmHg | -6.7 (14.4)

12. Other Pre Specified Outcome: 24hr Ambulatory Systolic BP Change
Description: as for outcome 10
Time Frame: Baseline to 24 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Artery Ablation
Number analyzed (Participants) | 43
mmHg | -13.2 (15.5)

13. Other Pre Specified Outcome: 24hr Ambulatory Diastolic BP Change
Description: as for outcome 10
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Artery Ablation
Number analyzed (Participants) | 44
mmHg | -5.7 (7.9)

14. Other Pre Specified Outcome: 24hr Ambulatory Diastolic BP Change
Description: as for outcome 10
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Artery Ablation
Number analyzed (Participants) | 35
mmHg | -4.3 (8.2)

15. Other Pre Specified Outcome: 24hr Ambulatory Diastolic BP Change
Description: as for outcome 10
Time Frame: Baseline to 24 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Artery Ablation
Number analyzed (Participants) | 43
mmHg | -7.5 (8.8)

16. Other Pre Specified Outcome: Urine Albumin to Creatinine Ratio
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mg/g
Arm/Group | Renal Artery Ablation
Number analyzed (Participants) | 46
mg/g | 167.6 (493)

17. Other Pre Specified Outcome: Urine Albumin to Creatinine Ratio
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/g
Arm/Group | Renal Artery Ablation
Number analyzed (Participants) | 45
mg/g | 153.0 (454)

18. Other Pre Specified Outcome: Urine Albumin to Creatinine Ratio
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mg/g
Arm/Group | Renal Artery Ablation
Number analyzed (Participants) | 45
mg/g | 116.9 (421)

19. Other Pre Specified Outcome: Urine Albumin to Creatinine Ratio
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: mg/g
Arm/Group | Renal Artery Ablation
Number analyzed (Participants) | 44
mg/g | 131.0 (358)

20. Other Pre Specified Outcome: Urine Albumin to Creatinine Ratio
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: mg/g
Arm/Group | Renal Artery Ablation
Number analyzed (Participants) | 44
mg/g | 157.5 (609)

21. Other Pre Specified Outcome: Estimated Glomular Filtration Rate
Description: Calculated using Modifide Diet in Renal Disease formula.
  estimated GFR = 186 x SerumCr-1.154 * age-0.203 * 1.212 (if patient is black) * 0.742 (if female)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mL/min per 1.73m^2
Arm/Group | Renal Artery Ablation
Number analyzed (Participants) | 46
mL/min per 1.73m^2 | 84.7 (18.0)

22. Other Pre Specified Outcome: Estimated Glomular Filtration Rate
Description: as for outcome 21
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mL/min per 1.73m^2
Arm/Group | Renal Artery Ablation
Number analyzed (Participants) | 45
mL/min per 1.73m^2 | 79.8 (19.5)

23. Other Pre Specified Outcome: Estimated Glomular Filtration Rate
Description: as for outcome 21
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mL/min per 1.73m^2
Arm/Group | Renal Artery Ablation
Number analyzed (Participants) | 45
mL/min per 1.73m^2 | 84.2 (20.3)

24. Other Pre Specified Outcome: Estimated Glomular Filtration Rate
Description: as for outcome 21
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: mL/min per 1.73m^2
Arm/Group | Renal Artery Ablation
Number analyzed (Participants) | 44
mL/min per 1.73m^2 | 75.5 (18.6)

25. Other Pre Specified Outcome: Estimated Glomular Filtration Rate
Description: as for outcome 21
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: mL/min per 1.73m^2
Arm/Group | Renal Artery Ablation
Number analyzed (Participants) | 44
mL/min per 1.73m^2 | 76.4 (25.3)

26. Other Pre Specified Outcome: Cystatin C
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Renal Artery Ablation
Number analyzed (Participants) | 46
mg/L | 1.1 (0.3)

27. Other Pre Specified Outcome: Cystatin C
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Renal Artery Ablation
Number analyzed (Participants) | 45
mg/L | 1.0 (0.2)

28. Other Pre Specified Outcome: Cystatin C
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Renal Artery Ablation
Number analyzed (Participants) | 45
mg/L | 0.9 (0.2)

29. Other Pre Specified Outcome: Cystatin C
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Renal Artery Ablation
Number analyzed (Participants) | 44
mg/L | 1.1 (0.3)

30. Other Pre Specified Outcome: Cystatin C
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Renal Artery Ablation
Number analyzed (Participants) | 44
mg/L | 1.3 (0.4)

ADVERSE EVENTS:
Time Frame: 24 months
Description: Events adjudicated by an independent clinical events committee.
Arm/Group | Renal Artery Ablation
Serious Adverse Events (participants affected / at risk) | 14/46
Other Adverse Events (participants affected / at risk) | 32/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Renal Artery Ablation (N=46)
Hypotension (Procedure Related) (General disorders) | 1 (1)
Hypertensive Renal Disease Progression (Device and Procedure Related) (Renal and urinary disorders) | 1 (1)
Renal Artery Stenosis (Device and Procedure Related) (Vascular disorders) | 1 (2)
ACCELERATED HYPERTENSION (Unrelated) (General disorders) | 1 (1)
ACUTE NSTEMI (Unrelated) (Cardiac disorders) | 1 (1)
ACUTE RENAL FAILURE (Unrelated) (Renal and urinary disorders) | 1 (1)
ATYPICAL CHEST PAIN (Unrelated) (General disorders) | 3 (3)
BACK PAIN (Unrelated) (General disorders) | 1 (1)
CEREBROVASCULAR ACCIDENT (Unrelated) (Vascular disorders) | 1 (1)
CLAUDICATION (Unrelated) (General disorders) | 1 (1)
GOUT (Unrelated) (Metabolism and nutrition disorders) | 1 (1)
HEADACHE (Unrelated) (General disorders) | 1 (1)
HEART FAILURE (Unrelated) (Cardiac disorders) | 1 (1)
HYPERTENSIVE RENAL DISEASE PROGRESSION (Unrelated) (General disorders) | 2 (2)
LEG TRAUMA (Unrelated) (Injury, poisoning and procedural complications) | 1 (1)
LEG WOUND CELLULITIS (Unrelated) (Infections and infestations) | 1 (1)
LUMBAR DISC DISEASE (Unrelated) (Musculoskeletal and connective tissue disorders) | 1 (1)
MELANOMA (Unrelated) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
METASTATIC CANCER (Unrelated) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
PANCREATITIS (Unrelated) (General disorders) | 1 (1)
VIRAL ILLNESS (Unrelated) (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Renal Artery Ablation (N=46)
BRADYCARDIA (Procedure Related) (Cardiac disorders) | 2 (2)
HEMATOMA (Procedure Related) (Blood and lymphatic system disorders) | 7 (7)
HYPOTENSION (Procedure Related) (General disorders) | 3 (3)
NAUSEA/VOMITING (Procedure Related) (Gastrointestinal disorders) | 1 (1)
PAIN (Procedure Related) (General disorders) | 2 (2)
VASOVAGAL RESPONSE (Procedure Related) (General disorders) | 2 (3)
HEMATOMA (Device and Procedure Related) (Blood and lymphatic system disorders) | 1 (1)
HYPERTENSIVE RENAL DISEASE PROGRESSION (Device and Procedure Related) (Renal and urinary disorders) | 1 (1)
PAIN (Device and Procedure Related) (General disorders) | 1 (1)
RENAL ARTERY STENOSIS (Device and Procedure Related) (Vascular disorders) | 1 (1)
TRANSIENT HEMATURIA/DISCOLORED URINE (Device and Procedure Related) (Renal and urinary disorders) | 1 (1)
VASOSPASM (Device and Procedure Related) (Vascular disorders) | 7 (12)
ALLERGIC REACTION (Unrelated) (Immune system disorders) | 1 (2)
ARM TREMOR (Unrelated) (General disorders) | 1 (1)
BACK PAIN (Unrelated) (General disorders) | 1 (1)
BROKEN FINGERS (Unrelated) (Injury, poisoning and procedural complications) | 1 (1)
DIABETES (Unrelated) (Metabolism and nutrition disorders) | 1 (1)
DIZZINESS (Unrelated) (General disorders) | 2 (2)
EDEMA (Unrelated) (General disorders) | 1 (1)
FIRST DEGREE AV BLOCK (Unrelated) (Cardiac disorders) | 1 (1)
HEADACHE (Unrelated) (General disorders) | 3 (4)
HYPERKALEMIA (Unrelated) (General disorders) | 1 (1)
HYPERTENSIVE HEADACHES (Unrelated) (General disorders) | 1 (1)
HYPERTENSIVE RELATED HEART FAILURE (Unrelated) (Cardiac disorders) | 1 (1)
HYPERTENSIVE RENAL DISEASE PROGRESSION (Unrelated) (Renal and urinary disorders) | 2 (2)
HYPOKALEMIA (Unrelated) (General disorders) | 2 (2)
HYPOTENSION (Unrelated) (General disorders) | 2 (2)
INFECTION (Unrelated) (Infections and infestations) | 4 (5)
PAIN (Unrelated) (General disorders) | 2 (2)
PARA-AORTIC LYMPADENOPATHY (Unrelated) (General disorders) | 1 (1)
PNEUMONIA (Unrelated) (Infections and infestations) | 1 (1)
PROTEINURIA (Unrelated) (Renal and urinary disorders) | 1 (1)
SKIN CANCER (Unrelated) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
SUPRAVENTRUCULAR TACHYCARDIA (Unrelated) (Cardiac disorders) | 1 (1)
TONSILLITIS (Unrelated) (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less